CLINICAL TRIAL: NCT02012101
Title: The Efficacy of Non-invasive Mechanical Ventilation as a Rescue Therapy for Relieving Dyspnea in Patients With Stable Severe COPD
Brief Title: Non-invasive Mechanical Ventilation as a Rescue Therapy to Relieve Dyspnea in Patients With Stable Severe COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yonger Ou, MMSc, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009CB522111
Record Dates: First submitted 2013-12-08; First posted 2013-12-16 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; dyspnea; exercise; Noninvasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity | interventions — Noninvasive Ventilation; Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- niv plus oxygen therapy (Experimental): oxygen therapy is given during the whole experimental process, niv is given at peak exercise until the borg scale reaches it's baseline point
  Interventions: Device: niv plus oxygen therapy
- oxygen therapy (Active Comparator): oxygen therapy is given during the whole experimental process
  Interventions: Device: oxygen therapy

INTERVENTIONS:
Device: niv plus oxygen therapy — NIV given on Philips Respironics BiPAP Vision apparatus.
  Other Names: Philips Respironics BiPAP Vision
  Arms: niv plus oxygen therapy
Device: oxygen therapy
  Arms: oxygen therapy

SUMMARY:
The purpose of this study is to determine whether non-invasive mechanical ventilation(NIV), playing the role as a rescue therapy , are effective in relieving exertional dyspnea in stable severe COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease(COPD) is a preventable and treatable illness, which is clinically characterized by persistent airflow limitation that is usually progressive. It's well known that airflow limitation lead to air trapping particularly during exercise, resulting in increased dyspnea and limitation of exercise capacity. Thus, COPD patients often unconsciously adopt a sedentary lifestyle, probably due to distressing exertional dyspnea. The sedentarism results in physical deconditioning and alterations of the peripheral muscles, and the latter one causes more exertional dyspnea and fatigue, which in turn leads to much more sedentarism, forming the vicious cycle of sedentarism, dyspnea/fatigue and more sedentarism. Thereby, measures should be taken to interrupt this vicious cycle. Some previous studies suggested that niv acting as an add-on therapy could help unloading the inspiratory muscle, reducing the dynamic compression of the airway, diminishing the dynamic hyperinflation,to some extent, relieved dyspnea during exercise in COPD patients. However,those measures were taken during exercise, acting as an add-on therapy. Whether NIV can play a role as a rescue therapy to relieve exertional dyspnea while the patients are already undergoing optimal treatment with bronchodilator and anti-inflammatory medication is still not quite clear. Therefore, we hypothesize that niv as a rescue-therapy has the same effect on relieving dyspnea in stable severe COPD patients just like the add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* severe COPD (post bronchodilator FEV1/FVC < 70% and FEV1 < 50% predicted)
* stable clinical condition(no exacerbation in the 4 weeks prior to study participation with no change in medications)
* dyspnea as a main symptom that limited daily activities

Exclusion Criteria:

* obvious pulmonary bullae demonstrated by chest CT scan or X-ray examination
* facial trauma/malformation; recent facial, upper airway or upper gastrointestinal tract surgery
* oxygen saturation(SpO2) < 88% at rest with a fraction of inspired oxygen(FiO2) ≥ 0.5
* systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg at rest
* unstable angina or a myocardial infarct in the previous four weeks
* resting sinus tachycardia ( > 120 beats/min)
* patients with musculoskeletal or neurological disorders
* patients who are unable to give informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Borg scale | baseline,repeated measurement for about ten minutes after intervention

SECONDARY OUTCOMES:
Inspiratory capacity(IC) | baseline,repeated measurement for about ten minutes after intervention
surface electromyography(sEMG) | baseline,repeated measurement for about ten minutes after intervention
respiratory parameters | baseline,repeated measurement for about ten minutes after intervention
  minute ventilation(VE); tidal volume(Vt); respiratory rate(RR); inspiratory time(Ti); total duty cycle(Ttot)
oxygen saturation(SpO2) | baseline,repeated measurement for about ten minutes after intervention
Heart Rate(HR) | baseline,repeated measurement for about ten minutes after intervention
the total recovery time | repeated measurement for about ten minutes after intervention
mouth pressure(Pmo) | baseline,repeated measurement for about ten minutes after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, M.D., Principal Investigator — Sate Key Laboratory of Respiratory Disease, First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- State Key Laboratory of Respiratory Disease, First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China